CLINICAL TRIAL: NCT05090124
Title: Experimental Medicine Studies of Brain and Peripheral Immune Mechanisms for Sickness Behaviours in Patients With Rheumatoid Arthritis
Brief Title: Experimental Medicine Studies of the Brain in Patients With Rheumatoid Arthritis REALISE
Acronym: REALISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GN18MH540
Record Dates: First submitted 2021-07-20; First posted 2021-10-22 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Sickness Behaviour; Tumour Necrosis Factor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Sodium Chloride; Injections

STUDY DESIGN:
Intervention Model Description: Participants will be randomised 1:1 to receive adalimumab or placebo. Upon exiting the study, those in the treatment arm will continue to receive adalimumab without delay and those in the placebo arm will begin adalimumab therapy under NHS standard of care.
Who Masked: Participant
Masking Description: This is a single-blind study, participants will be blinded to their study arm throughout.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-TNF treatment (Experimental): Adalimumab 40mg, will be administered as a subcutaneous injection once fortnightly on four occasions. No dose adjustments are permitted. The actual Adalimumab product selected at site will be dictated by what is used in standard care.
  The single-use, pre-filled syringe will be removed from storage at 2-8oC at least 30 minutes prior to administration to allow the contents to come to room temperature. The pre-filled syringe will be visually inspected for discolouration and particulates as per the product Summary of Product Characteristics.To facilitate maintenance of the blind, the pre-filled syringe (PFS) presentation will be used. The pen presentation will not be used.
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): Sodium chloride 0.9% for injection will be used as a placebo to adalimumab. An equal volume will be drawn up into a suitable sized syringe and labelled in accordance with standard practice at site. The dose will be administered as a subcutaneous injection once fortnightly on four occasions. No dose adjustments are permitted. Prior to administration, the prepared placebo syringe will be visually inspected for discolouration and particulate matter prior to administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab — Adalimumab 40mg, will be administered as a subcutaneous injection once fortnightly on four occasions. The actual Adalimumab product selected at site will be dictated by what is used in standard care.
  Other Names: Humira; Amgevita; Imraldi; Hyrimoz; Hulio
  Arms: anti-TNF treatment
Drug: Placebo — Sodium chloride 0.9% for injection will be used as a placebo. An equal volume will be drawn up into a suitable sized syringe and labelled in accordance with standard practice at site. The dose will be administered as a subcutaneous injection once fortnightly on four occasions.
  Other Names: Sodium chloride 0.9% for injection
  Arms: Placebo

SUMMARY:
The rationale for this study is to use immune molecule-specific drug treatment to leverage a mechanistic understanding of the brain changes that drive sickness behaviour. This will combine current therapy with innovative neuroimaging technologies to obtain data in humans that has hitherto only been available in animal studies. Data supporting the role of inflammatory molecules in sickness behaviours and other cognitive disorders are increasingly compelling. A putative mechanism linking inflammatory proteins to sickness behaviour is Tumour Necrosis Factor (TNF)-driven increases in extracellular glutamate leading to changes in neural function and brain network integrity and ultimately to sickness behaviour. Investigators hypothesise that TNF antagonism will effect changes in brain network connectivity and sickness behaviour score, that Rheumatoid Arthritis (RA) patients will show changes in brain network connectivity and glutamate quantification in the brain and that RA patients will show changes in monocyte infiltration into the brain that are correlated with changes in sickness behaviours. This is a randomised, placebo-controlled waiting list study. All patients will be eligible for anti-TNF treatment i.e. moderate to severe active disease as defined by Physician. Participants will be randomised to immediate (fast tracked) treatment or to treatment after 6-8 weeks (the routine waiting time). The latter group will receive placebo during the treatment phase.

DETAILED DESCRIPTION:
The study will involve participants aged over 18 years with RA and are scheduled to start outpatient anti-TNF treatment (with Adalimumab) as part of standard clinical care, who meet the inclusion criteria and none of the specified exclusion criteria. All will give full informed consent. This is a single-blind, randomised placebo-controlled waiting list study and after screening and consent, eligible participants will be randomised (1:1) to receive either adalimumab or placebo.

The study comprises standard care screening for anti-TNF therapy (incorporated into the study to allow us to fast track screening), a total of 7 research visits and one remote visit via telephone. At Visit 1 (Day 0) and Visit 4 ((14 ± 2 days from Visit 3), participants will undergo 7T MRI and MRS Neuroimaging protocols that incorporate resting-state and task-based fMRI and glutamate MRS measures. At Visit 1A (1 - 7 days from Visit 1) and Visit 4A (1 - 7 days from Visit 4), participants will undergo an optional SPECT scanning protocol. This visit will involve a 160ml blood draw, from which monocytes will be isolated and radiolabelled before being reinjected prior to SPECT scanning.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years < 75 years.
* Physician diagnosed moderate to severe RA.
* No previous biologic disease modifying antirheumatic drug therapy
* Usual care physician has confirmed the patient is eligible for anti-TNF treatment for active RA in line with the license for adalimumab (originator or biosimilar) and local practice subject to satisfactory completion of standard pre-biologic safety screening. Standard pre-biologic safety screening includes but not limited to exclusion of latent TB infection according to local protocol, chest X-ray, negative HIV screen, negative Hepatitis screen antibody, negative Hepatitis B surface antigen [Hep B sAg] and negative Hepatitis B anti-core antibody [Hep B cAb]

Note: Participant consent to treatment with adalimumab will have been obtained by the usual care team as per standard practice at site and will be prior to any approach for this study.

* Participant agrees to either immediate or delayed commencement of adalimumab.
* Self-reported sickness behaviour (fatigue, depression, anxiety) with one component > 4 on NRS
* Right-handed (to reduce neuroimaging heterogeneity).
* Women of Child-Bearing Potential (WoCBP) must be willing to use of effective contraception for study duration. Further information is provided in appendix 1
* Willing to participate and give informed consent for this research study.

Exclusion Criteria:

* Inability to provide written informed consent.
* Severe physical impairment (e.g. blindness, deafness, paraplegia).
* Pregnant, planning pregnancy or breast feeding.
* Serious infection including sepsis, tuberculosis and opportunistic infections such as invasive fungal infections.
* Severe liver or renal disease.
* Clinically diagnosed major confounding neurological disease including Multiple Sclerosis, Stroke, Traumatic Brain Injury, Parkinson's Disease, Alzheimer's Disease or similar neurodegenerative disease.
* Previous biologic disease modifying antirheumatic drug therapy with adalimumab, etanercept, qolimumab, infliximab, certolizumab, abatacept, tocilizumab, sarilumab, rituximab, tofacitinib or upadacitinib.
* Recent (within 4 weeks prior to Visit 1 baseline) use of intra-muscular or intra-articular steroid injections.
* Contraindications to MRI (e.g. metal implants, claustrophobia).
* Contraindications to Adalimumab.
* Concurrent or previous use of any other medicinal product (excluding vaccinations) that may, in the Principal Investigator's opinion, influence underlying disease activity through effects on immune and/or inflammatory responses.

If consenting to SPECT component, the following exclusions apply:

* Haemoglobin less than 100g/L
* Contraindications to SPECT protocol (e.g. hypersensitivity to Technetium or Stannous Chloride, recent Nuclear Medicine Procedure)
* Unwilling not to donate body fluids such as blood, sperm etc. for at least 24 hours after SPECT imaging at visits 1A and 4A.
* Unwilling to avoid close contact with children or people who are pregnant for 24 hours following SPECT imaging

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Change in sickness score as measured using the sickness questionnaire | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  The sickness questionnaire is a 10-item instrument used to capture perceived sickness behaviour. It was developed to display sensitivity to an inflammatory challenge and have adequate psychometric properties.
Change in brain connectivity as measured by 7T MRI | Visit 1 (Baseline, Day 0) and Visit 4 (14 ± 2 days from Visit 3).
  Changes in dorsal attention network (DAN) - left inferior parietal lobule (LIPL) brain connectivity as measured by 7T MRI

SECONDARY OUTCOMES:
Changes in fatigue from Baseline to Visit 4 via BRAF Severity | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Fatigue, measured by BRAF severity
Changes in fatigue from Baseline to Visit 4 via PROMIS Fatigue | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Fatigue, measured by PROMIS-Fatigue.
Changes in Hyperalgesia from Baseline to Visit 4 via ACR-FM Scale | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Hyperalgesia, measured by the ACR-FM Scale (American College of Rheumatology Fibromyalgia Scale).
Changes in pain from Baseline to Visit 4 via McGill Pain Questionnaire | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Pain, measured by McGill Pain Questionnaire
Changes in pain from Baseline to Visit 4 via Michigan Body Map Regional Pain Intensity | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Pain, measured by Michigan Body Map Regional Pain Intensity.
Changes in pain from Baseline to Visit 4 via Finger Perception Task | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Pain, measured by Finger Perception Task.
Changes in pain from Baseline to Visit 4 via Neglect-like Symptoms Questionnaire. | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Pain, measured by Neglect-like Symptoms Questionnaire.
Changes in pain from Baseline to Visit 4 via Number Rating Scale - Pain | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Pain, measured by Number Rating Scale - Pain.
Changes in sleep disturbance from Baseline to Visit 4 | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Sleep disturbance, measured by PROMIS-Sleep related impairment.
Changes in mood from Baseline to Visit 4 via HADS | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Mood, measured by HADS (Hospital Anxiety Depression Scale).
Changes in mood from Baseline to Visit 4 via PROMIS-Depression | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Mood, measured by PROMIS-Depression
Changes in mood from Baseline to Visit 4 via PROMIS-Anxiety | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Mood, measured by PROMIS-Anxiety.
Changes in cognition from Baseline to Visit 4 | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Cognition, measured by Cognitive failures questionnaire.
Changes in processing speed from Baseline to Visit 4 | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Processing Speed, measured by Symbol Digit Modalities Test.
Changes in memory from Baseline to Visit 4 | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Memory, measured by Auditory Verbal Learning Test.
Changes in verbal fluency from Baseline to Visit 4 | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Memory, measured by Auditory Verbal Learning Test.
Change in brain network connectivity at Baseline and Visit 4 | Visit 1 (Baseline, Day 0) and Visit 4 (14 ± 2 days from Visit 3).
  Change in brain network connectivity as measured by 7T Magnetic Resonance Imaging (MRI).
Change in brain glutamate quantification at Baseline and Visit 4 | Visit 1 (Baseline, Day 0) and Visit 4 (14 ± 2 days from Visit 3).
  Change in brain glutamate quantification as measured by 7T Magnetic Resonance Spectroscopy (MRS).
Measures of RA disease activity from Baseline to Visit 4 via DAS28 | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Indices of of disease activity for Rheumatoid Arthritis as measured by DAS28 (Disease Activity Score-28).
Measures of RA disease activity from Baseline to Visit 4 via CDAI | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Indices of of disease activity for Rheumatoid Arthritis as measured by CDAI (Clinical Disease Activity Index).
Measures of RA disease activity from Baseline to Visit 4 via SDAI | Visit 1 (Baseline, Day 0), Visit 2 (14 ± 2 days from Visit 1 or Visit 1A), Visit 3 (14 ± 2 days from Visit 2), and Visit 4 (14 ± 2 days from Visit 3).
  Indices of of disease activity for Rheumatoid Arthritis as measured by SDAI (Simple Disease Activity Index).

OTHER OUTCOMES:
Changes in monocyte infiltration into the brain measured using SPECT | Visit 1A (1-7 days from Visit 1 Baseline, Day 0) and Visit 4A (1-7 days from Visit 4).
  Monocyte infiltration is measured using SPECT (Single-Photon Emission Computerized Tomography) at visits 1A (pre-treatment) and 4A (final visit for those consenting to SPECT).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cavanagh, MD, PhD, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Addenbrooks Hopsital, Cambridge
  - Neil Basu, Glasgow

IPD SHARING:
Plan to Share IPD: No